CLINICAL TRIAL: NCT06590961
Title: A Phase Ia/Ib, Open-label, Dose-escalation, and Dose-expansion Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamic of UBX-303061 in Subjects With Relapsed/Refractory B-Cell Malignancies
Brief Title: UBX-303061 in Subjects With Relapsed/Refractory B-Cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ubix Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UBX-303-101
Record Dates: First submitted 2024-08-27; First posted 2024-09-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/Refractory B-cell Malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: Phase 1a: Dose escalation study Phase 1b: Dose expansion study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UBX-303061 (Experimental): UBX-303061
  Interventions: Drug: UBX-303061

INTERVENTIONS:
Drug: UBX-303061 — UBX-303061 oral dosage

SUMMARY:
This is a first-in-human Phase 1a/1b multicenter, open-label study designed to evaluate the safety and anti-cancer activity of UBX-303061 in patients with relapsed/refractory B-cell malignancies.

ELIGIBILITY:
Key Inclusion Criteria

* Capable of giving signed informed consent
* Age ≥18 years
* ECOG performance status ≤2.
* Phase Ia (dose-escalation part only): Subjects with relapsed and/or refractory B-cell malignancies (CLL/SLL, DLBCL, FL, MCL, WM or MZL) who have received at least 2 prior therapies and for subjects with no available treatment options as per the Investigator's discretion.
* Phase Ib (dose-expansion only): Subjects with relapsed and/or refractory B-cell malignancies who have received at least 2 prior therapies and for subjects with no available treatment options as per the Investigator's discretion, and fit into one of the following groups: CLL/SLL or DLBCL or MCL or FL, WM, MZL
* All subjects must have evaluable or measurable disease based on the appropriate tumor type criteria
* Adequate organ and bone marrow function

Key Exclusion Criteria

* For subjects with lymphoma:

  * Systemic antineoplastic therapy or any experimental therapy within 3 weeks or 5 half-lives, whichever is shorter, before the first dose of study treatment.
  * Therapy with tyrosine kinase inhibitor within 5 half-lives before the first dose of study treatment.
  * Unconjugated monoclonal antibody therapies <6 weeks before the first dose of study treatment.
  * Subjects that have undergone autologous stem cell rescue within 100 days prior to the first dose of study treatment.
  * Subjects that have undergone allogeneic stem cell transplant within 6 months prior to the first dose of study treatment.
  * Subjects with active graft-versus-host disease (GVHD) or on anti-GVHD treatment or prophylaxis.
  * History of chimeric antigen receptor T cell (CAR-T) therapy within 100 days prior to start of study drug.
  * Any immunotherapy within 4 weeks of first dose of study drug.
  * The time from the last dose of the most recent chemotherapy or experimental therapy to the first dose of study drug is <5 times the t1/2 of the previously administered agent(s).
* Previously exposed to BTK degradation therapy
* Malignant disease, other than that being treated in this study.
* Radiotherapy within 2 weeks of the first dose of study treatment
* Known hypersensitivity to BTK degraders or any of the ingredients.
* Impaired cardiac function or clinically significant cardiac disease
* Subjects with history of severe bleeding disorders and known/suspected other autoimmune disease
* Major surgery within 4 weeks of the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Protocol Specified Dose-Limiting Toxicities | 28-days
  Phase 1a and 1b
To establish the maximum tolerated dose and/or recommended Phase 1b dose(s) | Up to End of Treatment (up to 9 months)
  Phase 1a and 1b
Number of subjects with dose interruptions, reductions, and doses administered | Up to End of Treatment (up to 9 months)
  Phase 1a and qb

SECONDARY OUTCOMES:
To evaluate the anti-tumor activity of UBX-303061 in the dose levels based on Best overall response | Up to End of Treatment (up to 9 months)
  Phase 1a and 1b
To assess genetic markers including but not limited to BTK, PLCG2, MYD88 | Up to End of Treatment (up to 9 months)
  Phase 1a and 1b
To assess Cmin | 28-days
  Phase 1a and 1b
To assess tmax | 28-days
  Phase 1a and 1b
To assess AUC | 28-days
  Phase 1a and 1b
To assess Cmax | 28-days
  Phase 1a and 1b

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - Gabrail Cancer Center, Canton, Oklahoma
  - MD Anderson Cancer Center, Houston, Texas
- Poland (4):
  - MICS Centrum Medyczne Toruń, Torun, Kuyavian-Pomeranian Voivodeship
  - Pratia, MTZ Clinical Research, Warsaw, Mazowieckie Voivodeship
  - Pratia, Oncology Katowice, Katowice, Silesian Voivodeship
  - AidPort, Grodzisk Wielkopolski, Wielkopolskie Voivodeship
- South Korea (4):
  - Asan Medical Center, Seoul, Seoul
  - Samsung Medical Center, Seoul, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: No